CLINICAL TRIAL: NCT00917709
Title: In Vivo SPECT Imaging of Vesicular Acetylcholine and Dopamine Transporters in Dementia With Lewy Bodies: Applying in Diagnostic and Identification of Pathological Subtypes.
Brief Title: Imaging of Vesicular Acetylcholine and Dopamine Transporters in Dementia With Lewy Bodies
Acronym: IBVM/DATSCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHUBX 2008/34
Record Dates: First submitted 2009-06-05; First posted 2009-06-10 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Dementia With Lewy Bodies
Keywords: dementia with Lewy bodies; imaging; acetylcholine; dopamine; IBVM; DATSCAN
MeSH Terms: conditions — Lewy Body Disease | interventions — X-Rays; ioflupane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DLB with extrapyramidal syndrome (Experimental): patients dementia with Lewy bodies with extrapyramidal syndrome
  Interventions: Other: Imaging with IBVM; Other: Imaging with DATSCAN; Behavioral: neuropsychological evaluation
- DLB without extrapyramidal syndrome (Other): patients dementia with Lewy bodies without extrapyramidal syndrome
  Interventions: Other: Imaging with IBVM; Other: Imaging with DATSCAN; Behavioral: neuropsychological evaluation
- healthy volunteers (Sham Comparator): healthy volunteers
  Interventions: Other: Imaging with IBVM; Other: Imaging with DATSCAN; Behavioral: neuropsychological evaluation

INTERVENTIONS:
Other: Imaging with IBVM — in vivo molecular imaging of presynaptic molecular target of cholinergic systems with [123I]-iodobenzovesamicol
Other: Imaging with DATSCAN — in vivo molecular imaging of presynaptic molecular target of dopaminergic systems (DAT) with DATSCAN
Behavioral: neuropsychological evaluation — neuropsychological evaluation using neuropsychological tests

SUMMARY:
The general aim of this research project is to determine the relationships between alterations of central cholinergic (ACh) and dopaminergic (DA) systems and neurobehavioral features of dementias with Lewy bodies (DLB).

Both clinical and neurochemical data support the view that DLB is not a homogeneous entity and it can be hypothesized that differential alterations of central ACh systems (i.e. anterior vs posterior vs striatal interneurons) in association or not with a DA nigrostriatal dysfunction could partly support the clinical heterogeneity observed in this disease. ACh in vivo imaging has been relatively underutilized to date and to our knowledge only on the postsynaptic side. Furthermore, ACh/DA interactions and their relationships with the symptomatology of DLB and related pathologies (PDD) had never been investigated.

DETAILED DESCRIPTION:
Neurochemical investigations and observations suggest a crucial physiopathological role of central ACh systems in dementias with Lewy bodies (DLB). Alterations of cholinergic neurons could be involved in the general cognitive decline (central feature) but also in fluctuating attentional performances and rapid eye movement sleep disorder as it was shown in thalamus.

Post synaptic in vivo SPECT imaging recently demonstrated an increase in muscarinic receptors in DLB patients in the occipital cortex that could be associated with the visuospatial dysfunction often reported in DLB or even in visual hallucinations.From a pharmacological point of view, the involvement of ACh systems in DLB is confirmed by the consistently reported efficacy of cholinesterase inhibitor therapy, considered as greater than in AD.

Concerning DA systems, presynaptic in vivo SPECT imaging studies of DA transporter have shown a decreased striatal uptake in DLB patients, different when compared with Parkinson's disease patients or Alzheimer's disease patients.

Strategy, procedure In this project we will use for the first time in vivo molecular imaging of presynaptic molecular target of ACh systems (VAChT) with [123I]-iodobenzovesamicol and of DA systems (DAT) with DATSCAN in order to better analyse the link between neurobehavioral profiles of patients and a differential alteration of ACh/DA systems in DLB.

ELIGIBILITY:
Inclusion Criteria:

* Patients: man or woman probable DLB, with and without extrapyramida syndrome
* Healthy subjects: man or woman with no neuropsychiatric disorders

Exclusion Criteria:

* Diagnostic or therapeutic irradiation during the 12 months before SPECT imaging
* Age less than 18 and more than 90
* Iodine sensibility
* Brain-vascular disease, severe brain injury, type I and II diabetes mellitus, thyroid dysfunction, chronic alcoholism
* Pregnant and breast feeding women, women in age to procreate
* Impossibility to undergo MRI study (pace-maker, claustrophobia)
* Persons under guardianship, outside state to express their assent or in emergency situation
* Healthy subjects: cognitive impairment, dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Binding Potential (BP) quantification of each radioligand | Day 1 ; Day 1 and between day 14 to 28

SECONDARY OUTCOMES:
Ratio dopaminergic system/cholinergic system Binding Potential | Day 1 and between day 14 to 28

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Groupe Hospitalier Pellegrin - C.H.U. de Bordeaux, Bordeaux, France